CLINICAL TRIAL: NCT07017114
Title: Phase I, Dose-Escalation Clinical Trial to Evaluate the Safety and Tolerability of Pentoxifylline PKB171 Gel in Single-Dose Intravaginal Administration, Followed by an Extension Study With Multiple-Dose Administration in Healthy Volunteers
Brief Title: Pentoxifylline PKB171 Gel in Healthy Females Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Prokrea BCN, S.L. (Industry)
Collaborators: TFS Trial Form Support (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: PKB171-01; 2015-004611-21 (EudraCT Number)
Record Dates: First submitted 2025-01-28; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Safety; Pharmacokinetics; Maximum Tolerated Dose
Keywords: Pharmacokinetics; Maximum tolerated dose (MTD); Local tolerability; pentoxifyline PKB171 Gel

STUDY DESIGN:
Intervention Model Description: Dose-Escalation:
  A single dose of PKB171 vaginal gel (5 g) was intravaginally administered to healthy volunteers. Three strengths of PKB171 gel were tested: 2% (100 mg), 3% (150 mg) and 4% (200 mg).
  Three cohorts of 8 healthy female volunteers participated. For each dose level, subjects were randomly allocated to receive either the study drug or the placebo (3:1) between day 7 and 21 of their menstrual cycle.
  Safety and tolerability of each strength level and dose-escalation decisions. Full PK profile of PKB171 at each dose, blood samples (10 ml) were collected at baseline (pre-treatment), 10 minutes, 20 minutes, 30 minutes, 45 minutes, 1 h, 2 h, 4 h, 8 h and 24 hours post-adm were made based on the occurrence of drug-related adverse events (AEs).
  Multiple-dose extension substudy:
  The extension substudy was planned in order to assess the tolerability and PK of PKB171 after multiple-dose administration (two consecutive days) using the MTD in healthy female volunteers.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- PKB vaginal gel, at 100 mg pentoxifyline (2% gel). (Experimental): Regarding the dosing schedule, on day 1 of the study (Visit 1) a single dose of investigational drug (of each concentration) or placebo, were administered by intravaginal via using an applicator device (syringe).
  Interventions: Drug: Gel PKB171; Drug: Gel PKB171 placebo
- PKB vaginal gel, at 150 mg pentoxifyline (3% gel). (Experimental): Regarding the dosing schedule, on day 1 of the study (Visit 1) a single dose of investigational drug (of each concentration) or placebo, were administered by intravaginal via using an applicator device (syringe).
  Interventions: Drug: Gel PKB171; Drug: Gel PKB171 placebo
- PKB vaginal gel, at 200 mg pentoxifyline (4% gel). (Experimental): Regarding the dosing schedule, on day 1 of the study (Visit 1) a single dose of investigational drug (of each concentration) or placebo, were administered by intravaginal via using an applicator device (syringe).
  Interventions: Drug: Gel PKB171; Drug: Gel PKB171 placebo
- Placebo for PKB171 (Experimental): Placebo for PKB171 in Part A: dose-escalation and Part B: multiple-dose extension substudy
  Interventions: Drug: Gel PKB171; Drug: Gel PKB171 placebo

INTERVENTIONS:
Drug: Gel PKB171 — Subjects received a single dose of pentoxifylline PKB171 gel or placebo, in a one-dose form with an applicator device that allowed for vaginal administration following the randomisation list:
  * First dose level: 2% (100 mg)
  * Second dose level: 3% (150 mg)
  * Third dose level: 4% (200 mg) The treatment was provided by a member of the investigator's staff and self-administered by volunteers under clinical supervision.
  The dose-escalation process enabled to determine MTD or the highest dose that was safe to administer in later studies was determined. The results of this study helped to define the recommended doses to be used in the multiple-dose extension.
  Other Names: pentoxifyline gel
Drug: Gel PKB171 placebo — PKB vaginal gel at the MTD or placebo once every 24 hours for two consecutive days
  Other Names: placebo gel

SUMMARY:
A Phase I, Randomised, Double-Blind, Placebo-Controlled, Dose-Escalation Clinical Trial to evaluate the Safety and Tolerability of Pentoxifylline PKB171 Gel in Single-Dose Intravaginal Administration, followed by an Extension Study with Multiple-Dose Administration in Healthy Volunteers. The primary ojective was to determine the maximum tolerated dose (MTD) in terms of local tolerability of PKB171 after single-dose intravaginal administration in healthy female volunteers; the secondary objectives evaluated the safety and tolerability of PKB171 after single-dose intravaginal administration and the pharmacokinetic (PK) profile of PKB171 after single-dose intravaginal administration.

The extension substudy evaluated the safety and tolerability of PKB171 after multiple-dose intravaginal administration at the MTD in healthy volunteers.

DETAILED DESCRIPTION:
Phase I, randomised, double-blind, placebo-controlled, dose-escalation study to determine the MTD of PKB171 after single-dose intravaginal administration, followed by a double-blind extension study with multiple-dose vaginal administration (two consecutive days) of PKB171at the MTD in healthy volunteers.

Part A. Dose-Escalation:

A single dose of PKB171 vaginal gel (5 g) was intravaginally administered to healthy volunteers. Three strengths of PKB171 gel were tested: 2% (100 mg pentoxifyline), 3% (150 mg pentoxifyline) and 4% (200 mg pentoxifyline).

Three cohorts of 8 healthy female volunteers participated. Intrapatient dose escalation was not permitted. For each dose level, subjects were randomly allocated to receive either the study drug or the placebo (3:1) between day 7 and 21 of their menstrual cycle. In the first cohort (cohort A), a first volunteer received the study drug; after 24 hours of safety assessment, the rest of the volunteers of that cohort received the study drug (5 volunteers) or placebo (2 volunteers).

Safety and tolerability of each strength level and dose-escalation decisions were made based on the occurrence of drug-related adverse events (AEs). The maximum tolerated dose (MTD) in terms of local tolerability was defined as the highest dose at which no more than 1 of 6 patients experienced a moderate or severe drug-related adverse events following PKB171 gel administration. Dose escalation proceeded until the highest strength of PKB171 vaginal gel (4%) or matching placebo.

To obtain a full PK profile of PKB171 at each dose, blood samples (10 ml) were collected at baseline (pre-treatment), 10 minutes, 20 minutes, 30 minutes, 45 minutes, 1 h, 2 h, 4 h, 8 h and 24 hours post-administration (10 blood draws in total) to analyse the pharmacokinetic parameters (Cmax, Tmax, AUC0-t, T1/2, Vd, Clp) of PKB171 and its metabolite 5-OH-pentoxifylline.

Part B. Multiple-dose extension substudy:

After completing the dose-escalation phase, an extension substudy was planned in order to assess the tolerability and PK of PKB171 after multiple-dose administration (two consecutive days) using the MTD in healthy female volunteers.

A subgroup of 6 patients that have participated in the first part of the study were invited to participate in the randomised, parallel-group, placebo-controlled extension study. Patients were randomly allocated to receive either the study drug or the placebo (2:1) between day 7 and 21 of their menstrual cycle. The MTD of PKB171 gel or matching placebo (5 g) were administered intravaginally in two consecutive days.

ELIGIBILITY:
Inclusion criteria

Subjects had to fulfil all the following criteria to be eligible for study entry:

1. Understand and agree to the trial procedures and sign an informed consent form.
2. Female volunteers aged between 18 and 45 years.
3. Regular menstrual cycle (regardless of menstrual cycle length)*

   *Subjects were asked for the duration of their menstrual cycle and the date of last menstruation in order to identify the stage of their menstrual cycle between days 7 and 21, and depending on their menstrual cycle they were distributed over the three consecutive study periods (and also to have them identified for the extension substudy).
4. Medical records and physical examination showing no organic or psychiatric disorders.
5. Gynaecological examination with visual inspection by the gynaecologist to rule out possible signs/symptoms of inflammation or vaginal infection and/or other gynaecological diseases, such as vulvovaginitis, infectious vulvovaginitis, candidal vulvovaginitis or fungal infection, trichomoniasis, bacterial vaginosis, irritative vulvovaginitis (due to the use of vaginal douching, deodorants, etc.), condylomata or genital warts, bartholinitis, cervicitis, etc. Symptoms: increased vaginal discharge and characteristics' change (colour, smell, texture and appearance) that varied according to the agent causing the infection, redness of the vulvar and vaginal mucosae, warts on the labia and/or anus, painful lump (with abscess), etc.

   In addition, during clinical examination, the gynaecologist asked volunteers about the presence of symptoms (pruritus or itching of the external genitalia and/or vagina, sensation of burning or stinging in the genitalia, urinary tract problems such as frequent urination, burning urination, heavy flow, etc.) to confirm the diagnosis.
6. ECG, vital signs and blood and urine tests performed prior to the trial had to be within normal limits. Minor or one-off variations from the normal limits were allowed at the principal investigator's discretion, insofar as they do not pose a risk to subjects and do not interfere in the evaluation of the drug.
7. Body mass index (BMI=weight/height2) should be between 18.5 and 24.99 kg/m2
8. Women who have not participated in a clinical trial involving drugs in the three months prior to this study.

DIAGNOSIS AND MAIN CRITERIA FOR INCLUSION:

Inclusion criteria

Subjects had to fulfil all the following criteria to be eligible for study entry:

1. Understand and agree to the trial procedures and sign an informed consent form.
2. Female volunteers aged between 18 and 45 years.
3. Regular menstrual cycle (regardless of menstrual cycle length)*

   *Subjects were asked for the duration of their menstrual cycle and the date of last menstruation in order to identify the stage of their menstrual cycle between days 7 and 21, and depending on their menstrual cycle they were distributed over the three consecutive study periods (and also to have them identified for the extension substudy).
4. Medical records and physical examination showing no organic or psychiatric disorders.
5. Gynaecological examination with visual inspection by the gynaecologist to rule out possible signs/symptoms of inflammation or vaginal infection and/or other gynaecological diseases, such as vulvovaginitis, infectious vulvovaginitis, candidal vulvovaginitis or fungal infection, trichomoniasis, bacterial vaginosis, irritative vulvovaginitis (due to the use of vaginal douching, deodorants, etc.), condylomata or genital warts, bartholinitis, cervicitis, etc. Symptoms: increased vaginal discharge and characteristics' change (colour, smell, texture and appearance) that varied according to the agent causing the infection, redness of the vulvar and vaginal mucosae, warts on the labia and/or anus, painful lump (with abscess), etc.

   In addition, during clinical examination, the gynaecologist asked volunteers about the presence of symptoms (pruritus or itching of the external genitalia and/or vagina, sensation of burning or stinging in the genitalia, urinary tract problems such as frequent urination, burning urination, heavy flow, etc.) to confirm the diagnosis.
6. ECG, vital signs and blood and urine tests performed prior to the trial had to be within normal limits. Minor or one-off variations from the normal limits were allowed at the principal investigator's discretion, insofar as they do not pose a risk to subjects and do not interfere in the evaluation of the drug.
7. Body mass index (BMI=weight/height2) should be between 18.5 and 24.99 kg/m2
8. Women who have not participated in a clinical trial involving drugs in the three months prior to this study.

Exclusion criteria

Subjects who met any of the following conditions were not selected for this trial:

1. Subjects who were not able to understand the nature of the trial and the procedures that they were asked to follow.
2. History or clinical evidence of gastrointestinal, liver, renal or other types of disorders that led to a change in how the drug was absorbed, distributed, metabolised or excreted, or which suggested drug-induced gastrointestinal upset.
3. History or clinical evidence of psychiatric disorders, alcoholism, abuse of medication or other drugs, or habitual consumption of psychoactive drugs.
4. Any organic disease or major surgery in the 3 months prior to the start of the study.
5. Subjects who had intolerance or serious adverse reactions to the study drugs or any of their ingredients.
6. Regular use of medication in the month prior to the study sessions (including birth control or hormone therapy of any kind), except for vitamins or dietary supplements that, in the opinion of the principal investigator or designated supporting staff, involved no risk to subjects and did not interfere with the study objectives. In this case, subjects had to stop taking them from one week before the experimental sessions and until they had been completed. Treatment with single or limited symptomatic medication in the week prior to the study sessions was not cause for exclusion if it was calculated that it had been completely eliminated by the day of the experimental session.
7. Smoking more than 5 cigarettes a day.
8. Consuming more than 20 g of alcohol a day.
9. Subjects with positive serology for hepatitis B, C or HIV.
10. Women with a positive test for syphilis (RPR: rapid plasma reagin).
11. Pregnant or breast-feeding women.
12. Women who did not commit to using reliable birth control during the study
13. Women who had any contraindication specified in the summary of product characteristics of oral pentoxifylline.

To be eligible, subjects had to agree to the following restrictions regarding diet, sex, drug use and exercise during the study:

1. Did not perform any strenuous physical exercise in the 48 hours prior to the start of each session.
2. Did not take any type of drug from the screening visit to the end of the study.
3. Did not have intercourse relations with penetration in the 24 hours prior to the start of each study visit.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-01-27 (Actual); Primary Completion 2016-04-26 (Actual); Study Completion 2016-09-21 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of PKB171 | 3 weeks
  To determine the maximum tolerated dose (MTD) of PKB171 according to the dose at which a related adverse event occurs in one or more subjects.

SECONDARY OUTCOMES:
Adverse events | 3 weeks
  Evaluate the adverse events (AEs) reported spontaneusly by the subjects, as well as those what are evident to the investigator, including adverse reactions.
Local reactions of PKB171 | 3 weeks
  Evaluate local reactions observed by the gynaecoligist and/or reported by the volunteer after the treatment
Visual Analogue Scale | 3 weeks
  Evaluate the assessment of local reactions reported by VAS (Visual Analogue Scale). Is a straight horizontal line of fixed length, usually 100 mm. The ends are defined as the extreme limits of the parameter to be measured (symptom, pain, health) orientated from the left (worst) to the right (best)
Pregnancy | 3 weeks
  In case of pregnancy during the phase I study data collection, including information on pregnancy, fetal development and birth outcomes will be collected.
Peak Plasma Concentration (Cmax) | 3 weeks
  Complete PK profile at each concentration, blood samples (10mL) was drawn at baseline (pre-treatment), 10 minutes, 20 minutes, 30 minutes, 45 minutes, 1 h, 2 h, 4 h, 8 h and 12 h post-treatment (10 samples in total), in order to analyze the PK parameters of PKB171 and its metabolite 5-hydroxypentoxyphylline.
Tmax | 3 weeks
  Complete PK profile at each concentration, blood samples (10mL) was drawn at baseline (pre-treatment), 10 minutes, 20 minutes, 30 minutes, 45 minutes, 1 h, 2 h, 4 h, 8 h and 12 h post-treatment (10 samples in total), in order to analyze the PK parameters of PKB171 and its metabolite 5-hydroxypentoxyphylline.
Area Under the Curve (AUC0-t) | 3 weeks
  Complete PK profile at each concentration, blood samples (10mL) was drawn at baseline (pre-treatment), 10 minutes, 20 minutes, 30 minutes, 45 minutes, 1 h, 2 h, 4 h, 8 h and 12 h post-treatment (10 samples in total), in order to analyze the PK parameters of PKB171 and its metabolite 5-hydroxypentoxyphylline.
Volume of Distribution (Vd) | 3 weeks
  Complete PK profile at each concentration, blood samples (10mL) was drawn at baseline (pre-treatment), 10 minutes, 20 minutes, 30 minutes, 45 minutes, 1 h, 2 h, 4 h, 8 h and 12 h post-treatment (10 samples in total), in order to analyze the PK parameters of PKB171 and its metabolite 5-hydroxypentoxyphylline.
Half live (T1/2) | 3 weeks
  Complete PK profile at each concentration, blood samples (10mL) was drawn at baseline (pre-treatment), 10 minutes, 20 minutes, 30 minutes, 45 minutes, 1 h, 2 h, 4 h, 8 h and 12 h post-treatment (10 samples in total), in order to analyze the PK parameters of PKB171 and its metabolite 5-hydroxypentoxyphylline.
Blood test for pregnancy | 3 weeks
  A quantitative human chorionic gonadotropin (HCG or hCG) blood test measures the specific level of HCG in the blood. Results are given in milli-international units per milliliter (mIU/mL). In non-pregnant women is less than 5mIU/mL.
  In case of pregnancy during the phase I study data collection, including information on pregnancy, fetal development and birth outcomes will be collected.
Plasma Clearance (CLp) | 3 weeks
  Complete PK profile at each concentration, blood samples (10mL) was drawn at baseline (pre-treatment), 10 minutes, 20 minutes, 30 minutes, 45 minutes, 1 h, 2 h, 4 h, 8 h and 12 h post-treatment (10 samples in total), in order to analyze the PK parameters of PKB171 and its metabolite 5-hydroxypentoxyphylline.

CONTACTS AND LOCATIONS:
Overall Officials: José M Palacios, MD, Study Chair — ProkreaBCN, S.L.

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.